CLINICAL TRIAL: NCT00362856
Title: A Phase 2a, Randomized, Double-Blind, Placebo Controlled, Dose Ranging, Multicenter Study to Determine the Safety, Tolerance, and Efficacy of Larazotide Acetate (AT-1001) in Celiac Disease Subjects During Gluten Challenge.
Brief Title: Safety and Tolerability Study of Larazotide Acetate in Celiac Disease Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 9 Meters Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN1001-004
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Celiac Disease
Keywords: larazotide acetate
MeSH Terms: conditions — Celiac Disease | interventions — larazotide acetate

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo controlled, dose ranging, multicenter
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo + Gluten (Placebo Comparator): placebo TID + gluten 800 mg TID administered orally in capsules
  Interventions: Drug: Placebo
- Placebo + Gluten placebo (Placebo Comparator): placebo TID + gluten placebo TID administered orally in capsules
  Interventions: Drug: Placebo
- Larazotide acetate 8 mg + Gluten placebo (Other): Safety Control Arm. Larazotide acetate 8 mg TID + gluten placebo TID administered orally in capsules
  Interventions: Drug: larazotide acetate
- Larazotide acetate 0.25 mg + Gluten (Active Comparator): Larazotide acetate 0.25 mg TID + gluten 800 mg TID administered orally in capsules
  Interventions: Drug: larazotide acetate
- Larazotide acetate 1 mg + Gluten (Active Comparator): Larazotide acetate 1 mg TID + gluten 800 mg TID administered orally in capsules
  Interventions: Drug: larazotide acetate
- Larazotide acetate 4 mg + Gluten (Active Comparator): Larazotide acetate 4 mg TID + gluten 800 mg TID administered orally in capsules
  Interventions: Drug: larazotide acetate
- Larazotide acetate 8 mg + Gluten (Active Comparator): Larazotide acetate 8 mg TID + gluten 800 mg TID administered orally in capsules
  Interventions: Drug: larazotide acetate

INTERVENTIONS:
Drug: larazotide acetate — capsule
  Other Names: AT-1001; INN-202
  Arms: Larazotide acetate 0.25 mg + Gluten; Larazotide acetate 1 mg + Gluten; Larazotide acetate 4 mg + Gluten; Larazotide acetate 8 mg + Gluten; Larazotide acetate 8 mg + Gluten placebo
Drug: Placebo — capsule
  Arms: Placebo + Gluten; Placebo + Gluten placebo

SUMMARY:
This study was run to determine the safety, tolerance, and efficacy of multiple doses of larazotide acetate in subjects with celiac disease following a gluten challenge.

DETAILED DESCRIPTION:
CLIN1001-004 was a randomized, double-blind, placebo controlled, dose-ranging, 7-arm, multicenter study with a gluten challenge. The objects were multiple dose safety and tolerance; efficacy (intestinal permeability [change in urinary LAMA ratio] and disease signs and symptoms) following gluten challenge.

Following a 21-day screening period, subjects were randomized to one of seven treatments groups: four groups received larazotide acetate (0.25 mg, 1 mg, 4 mg or 8 mg TID) along with an 800 mg gluten challenge, one group received placebo with an 800 mg gluten challenge, a safety control arm received the highest dose of larazotide acetate (8 mg TID) and gluten placebo and the last group received drug placebo and gluten placebo. The gluten challenge was administered as capsules (800 mg TID) with each main meal for a total of 2.4 g daily. Drug or drug placebo was administered TID 15 minutes prior to each main meal. Subjects received their assigned treatments for two weeks (Day 0 through Day 14) and came to clinic for a follow-up visit one week later (Day 21). Subjects remained on their gluten-free diet for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have been diagnosed with celiac disease by biopsy for ≥ 6 months.
* Have a Anti-Tissue Transglutaminase (tTG) ≤ 10 EU as measured by serology.
* Must be on a gluten-free diet for at least the past 6 months.

Exclusion Criteria:

* Have any chronic active GI disease other than celiac disease (e.g., IBS, Crohn's, Colitis).
* Have diabetes (Type 1 or Type 2).
* Chronically consumes non-steroidal anti-inflammatory agents ("NSAIDs") or takes proton-pump inhibitors.
* Consuming oral corticosteroids or immune suppressants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-09-13 (Actual); Primary Completion 2007-03-06 (Actual); Study Completion 2007-03-06 (Actual)

PRIMARY OUTCOMES:
To demonstrate the safety and tolerability of multiple, oral doses of larazotide acetate in celiac disease subjects that maintain a gluten-free diet. | Safety measurements were performed at Screening and at Day 0, 7, 14, and 21 ('End of Study'). Any change from baseline value was calculated at each subsequent visit until "End of Study" (Day 21).
  Safety endpoints assessed in this study were adverse events, vital signs, hematology, clinical chemistry, urinalysis and ECG
To evaluate the efficacy of multiple dose levels of larazotide acetate in preventing intestinal permeability changes induced by gluten challenge | On Days 0, 6, 13, and 20 subjects drank a solution of lactulose and mannitol. Subject's urine was collected during the day on Day 0 and overnight prior to subsequent visits and analyzed for LAMA recoveries via standardized methodologies.
  The primary efficacy outcome was the Day 0-to-Day 14 change in urinary LAMA ratio ( a measure of intestinal permeability) as a response to gluten

SECONDARY OUTCOMES:
Changes in daily and weekly reported health outcomes | Symptom diary - daily; PGWBI - weekly; GSRS - weekly
  Health outcomes were assessed using a daily symptom diary; a weekly PGWBI and a weekly GSRS
Changes in urinary LAMA ratios between Day 0 to Day 7 | See Primary Outcome Measure No. 2
  See Primary Outcome Measure No. 2
Changes in urinary lactulose fractional excretion between Day 0 to Day 7 to Day 14 | See Primary Outcome Measure No. 2
  See Primary Outcome Measure No. 2
Changes in urinary mannitol fractional excretion between Day 0 to Day 7 to Day 14 | See Primary Outcome Measure No. 2
  See Primary Outcome Measure No. 2
Change in urinary nitrite / nitrate levels from Day 0 to Day 14 | Day 0 and Day 14
  Nitrite/nitrate levels were assessed for correlation to the measures of intestinal permeability
Change in anti-tTG levels from Screening to Day 21 | Screening and Day 21
  Changes between screening and Day 21 anti-tTG levels were assessed for correlation to the measures of intestinal permeability
Change in cell markers and cytokines from PBMCs | Days 0, 7, 14 and 21
  Serum cytokine and cell surface marker determinations were assessed for correlation to the measures of intestinal permeability
Changes in zonulin level | Days 0, 7, 14 and 21
  Serum zonulin levels were assessed for correlation to the measures of intestinal permeability

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Research Site, Scottsdale, Arizona
  - San Diego, California
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Morristown, New Jersey
  - Bismarck, North Dakota
  - Research Site, Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Research Site, Richmond, Virginia

REFERENCES:
- [Result] Leffler DA, Kelly CP, Abdallah HZ, Colatrella AM, Harris LA, Leon F, Arterburn LA, Paterson BM, Lan ZH, Murray JA. A randomized, double-blind study of larazotide acetate to prevent the activation of celiac disease during gluten challenge. Am J Gastroenterol. 2012 Oct;107(10):1554-62. doi: 10.1038/ajg.2012.211. Epub 2012 Jul 24. PMID 22825365